CLINICAL TRIAL: NCT02925273
Title: The Effect of Hand Grasping Techniques on Eliciting the Grasp Reflex in Patients With Dementia or Suspected Frontal Lobe Dysfunction
Brief Title: Hand Grasping Techniques on Eliciting the Grasp Reflex in Patients With Dementia
Acronym: GRASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Principal Investigator, Lauren Fedor, Program Manager, Rowan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GRASP
Record Dates: First submitted 2016-08-05; First posted 2016-10-05 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Dementia
Keywords: dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard (Other): Prospective, grasp techniques will be compared in each patient from the experimental group using a palmar grasp without dorsal stimulation and a standard palmar grasp test with dorsal stimulation on the same patient as the control group
  Interventions: Other: palmar grasp without dorsal stimulation; Other: standard palmar grasp test with dorsal stimulation

INTERVENTIONS:
Other: palmar grasp without dorsal stimulation — The patient will then be asked to keep the arms at 90 degrees and the researcher will slightly stroke palm and fingers of both hands of the patient simultaneously. After completion of each technique, the presence or absence of the response will be noted. In addition, the prominence of the response on the rating scale will be obtained as explained below.
  The scaling of the grasp response is as followed:
  1. Flexion at the distal interphalangeal joint of the hand
  2. Flexion at the proximal interphalangeal joint of the hand
  3. Flexion at the metacarpal-phalangeal joint of the hand
Other: standard palmar grasp test with dorsal stimulation — The patient will be asked to put their arms at 90 degrees and the researcher will hold one hand at the wrist and dorsum of the palm and lightly stroke the palm and fingers. The patient will be instructed to relax hands and not hold on while doing the grasp and see if the response persists. The same technique will be repeated for the patient's other hand.

SUMMARY:
In this study, the investigators will determine the difference between the two techniques used to elicit the grasp response in patients with frontal lobe dysfunction, primarily in dementia patients versus control patients.

DETAILED DESCRIPTION:
The goal of this project is to determine the optimal technique to elicit the grasping response in patients with dementia or suspected frontal lobe dysfunction. The proposed study is to perform two techniques to elicit grasp response in patients with dementia or suspected frontal lobe dysfunction and observe the presence or absence of the response and prominence of the response on a proposed rating scale. Future goals will be aimed at aiding clinicians in refining their clinical techniques to be more sensitive for diagnosing frontal lobe dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to sign informed consent or have a surrogate present to sign the consent
2. Age 18 or above
3. Patients are diagnosed with dementia, Alzheimer's disease, or frontal lobe dysfunction
4. Medications are to remain stable during the course of the study except for emergency modifications.

Exclusion Criteria:

1. Inability to obtain informed consent from patient or surrogate
2. Unable to follow commands.
3. Physical restrictions (i.e. spasticity of hands/arms, upper extremity amputation)
4. Other comorbidities such as muscular diseases, hepatic encephalopathy, renal failure, down syndrome, NPH, depression, and cerebral palsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07; Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Grasp response | six months
  The primary objective of the study will be to determine if a change in the performance of the grasp response will lead to a change in the way the response is elicited. The prominence of the grasp response will be scored on a rating scale

SECONDARY OUTCOMES:
Frontal Lobe release- Glabellar Response | six months
  The secondary objective during this study will be to determine if other frontal release signs are present in study participants. The glabellar response will be tested.
Frontal lobe release- Palmomental Response | six months
  The secondary objective during this study will be to determine if other frontal release signs are present in study participants. The palmomental response will be tested.
Frontal lobe release- Snout Response | six months
  The secondary objective during this study will be to determine if other frontal release signs are present in study participants. The snout response will be tested.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Barone, DO, Principal Investigator — Rowan University School of Osteopathic Medicine
Locations (1):
- Rowan University School of Osteopathic Medicine, Stratford, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No